CLINICAL TRIAL: NCT03374033
Title: Effect of High Protein and High Energy Intakes and Physical Activity on Growth and Body Composition of Extremely Low Birth Weight Infants: a Randomised Controlled Trial.
Brief Title: High Protein and High Energy Intakes and Physical Activity on Growth of Extremely Low Birth Weight Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, Head of Neonatology Department, Università Politecnica delle Marche
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DG-297
Record Dates: First submitted 2017-11-13; First posted 2017-12-15 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Preterm infants, growth, nutrition, physical activity
MeSH Terms: conditions — Motor Activity | interventions — NutR protein, bacteriophage lambda

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NUTR (Nutrition) 0_STIMUL(Stimulation) 0 (No Intervention): Standard Nutrition and no Physical Stimulation
- NUTR 0_STIMUL + (Experimental): Standard Nutrition and Physical Stimulation
  Interventions: Behavioral: STIMUL +
- NUTR +_STIMUL 0 (Experimental): Enhanced Nutrition, and no Physical Stimulation
  Interventions: Dietary Supplement: NUTR +
- NUTR +_STIMUL + (Experimental): Enhanced Nutrition and Physical Stimulation
  Interventions: Dietary Supplement: NUTR +; Behavioral: STIMUL +

INTERVENTIONS:
Dietary Supplement: NUTR + — one extra g/kg/d of protein and lipids starting before 48 hours after birth until 36 weeks postmenstrual age
  Arms: NUTR +_STIMUL +; NUTR +_STIMUL 0
Behavioral: STIMUL + — Physical activity stimulation consists in flexion/extension of the 4 limbs and other motion exercises of the shoulder girdle and of the hips. This stimulation will take place before the feed for a mean of 30 times a week (minimum 24- maximum 36 times a week, 10 minutes each time) and will start within the 10th day of life until 36 weeks postmenstrual age
  Arms: NUTR +_STIMUL +; NUTR 0_STIMUL +

SUMMARY:
The aim of this study is to evaluate the effect of increasing amino acid and energy intake during parenteral and enteral nutrition with and without the stimulation of the infant's physical activity, on growth of extremely low birth weight infants .

DETAILED DESCRIPTION:
Increasing protein and energy intake above the anabolic capacity of a given individual may result in increased lipogenesis and excessive fat deposition. Adults with reduced mobility or with neuromuscular conditions will develop excessive fat deposition if they receive normal to high protein and energy intakes. Excessive fat deposition have been demonstrated in preterm infants receiving high energy intakes. Given that physical activity in preterms is often reduced for the prematurity itself, the associated sickness and the numerous medications, the investigators speculate that physical stimulation may have a beneficial effect on protein accretion and on lean mass accretion. The investigators further hypothesize that today's recommended daily intakes of proteins and energy cannot be fully incorporated into lean body mass without a concomitant physical activity. In spite of the fact that this notion is well accepted in adult physiology and in the elderly, it has never been tested in preterm infants.

This factorial randomised controlled trial will evaluate the effect of increasing amino acid intake (by 1 g/kg/d) and energy intake (by 20 kcal/kg/d) during parenteral nutrition and also of increasing protein intake and energy intake by an extra 1 g/kg/d during enteral nutrition, with and without the stimulation of the infant's physical activity, on growth of extremely low birth weight infants. The investigators aim at demonstrating that increasing energy and protein intake above the standard of care intakes will result in better growth only in association with adequate physical activity, in particular in relation to body composition and lean mass accretion.

ELIGIBILITY:
Inclusion Criteria:

* 24 weeks < gestational age < 32 weeks
* inborn or outborn admitted before 24 hours of age
* parenteral or enteral nutrition start before 48 hours of age
* parental consent

Exclusion Criteria:

* difficulty in starting physical activity stimulation before 10 days of life
* death before 36 W PMA
* diagnosis of necrotising enterocolitis (before 36 W PMA)
* any major surgery (before 36 W PMA)
* congenital syndrome, severe malformations
* inborn errors of metabolism
* parental consent withdrawn

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-04-03 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Weight gain (Birth-36 Weeks PMA) | birth up to 36 weeks postmenstrual age
  Weight gain from birth up to 36 weeks postmenstrual age (g/kg/d)

SECONDARY OUTCOMES:
Muscle ultrasound | 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age(+-1d ), 36 weeks postmenstrual age(+-1d ), 40 weeks postmenstrual age(+-1d )
  Ultrasound measurement of mid thigh and mid arm muscle thickness (cm)
Adipose tissue ultrasound | 32 weeks postmenstrual age(+-1d ), 34 weeks postmenstrual age(+-1d ), 36 weeks postmenstrual age(+-1d ), 40 weeks postmenstrual age(+-1d )
  Ultrasound measurement of mid thigh and mid arm adipose tissue thickness (cm)
Lean body mass estimate using deuterium dilution | 36 weeks postmenstrual age (+-1d )
  Urinary deuterium enrichment after 6 and 12 hours from deuterium oral administration (baseline)
Skinfold thickness | 32 weeks postmenstrual age(+-1d ), 34 weeks postmenstrual age(+-1d ), 36 weeks postmenstrual age(+-1d ), 40 weeks postmenstrual age(+-1d ), between 22 and 24 months (2 years correct age)
  Biceps and triceps skinfold thickness (both arms) (cm)
Brain MRI | 40 weeks postmenstrual age (+-1d )
  Brain injury, growth and maturation according to Kidokoro et al.
Weight | birth, daily up to 36 weeks postmenstrual age; 40weeks postmenstrual age (+-1d ), between 22 and 24 months (2 years correct age)
  weight measured by a digital infant scale (g)
Total body length | birth, weekly until 36 weeks postmenstrual age; 40weeks postmenstrual age (+-1d ), between 22 and 24 months (2 years correct age)
  Total body length measured by a neonatal stadiometer (cm)
Head circumference | birth, weekly up to 36 weeks postmenstrual age; 40weeks postmenstrual age (+-1d ), between 22 and 24 months (2 years correct age)
  Head circumference measured by a flexible non-stretchable tape (cm)
Tibial length | birth, 32 weeks postmenstrual age(+-1d ), 34 weeks postmenstrual age(+-1d ), 36 weeks postmenstrual age(+-1d ), 40 weeks postmenstrual age(+-1d ), between 22 and 24 months (2 years correct age)
  Knee-heel length measured by knemometry (cm)
Weight gain (BW recovery-36W PMA) | birth weight recovery up to 36 weeks postmenstrual age
  Weight gain from the birth weight recovery until 36 weeks postmenstrual age (g/kg/d)
Bayley III Cognitive Score (MDI) | between 22 and 24 months (2 years correct age)
  Cognitive scale (range 55-145). The Scale has index mean scores of 100 (SD ± 15). An index composite score of < 70 (>2 SD below the mean) is defined to indicate severe impairment, while an index composite score of 70-84 (>1 SD below the mean) is defined to indicate mild impairment. Index composite scores ≥ 85 indicate normal development.
Bayley III Language Score | between 22 and 24 months (2 years correct age)
  Language scale (range 45-155). The Scale has index mean scores of 100 (SD ± 15). An index composite score of < 70 (>2 SD below the mean) is defined to indicate severe impairment, while an index composite score of 70-84 (>1 SD below the mean) is defined to indicate mild impairment. Index composite scores ≥ 85 indicate normal development.
Bayley III Motor Score (PDI) | between 22 and 24 months (2 years correct age)
  Motor scale (range 45-155). The Scale has index mean scores of 100 (SD ± 15). An index composite score of < 70 (>2 SD below the mean) is defined to indicate severe impairment, while an index composite score of 70-84 (>1 SD below the mean) is defined to indicate mild impairment. Index composite scores ≥ 85 indicate normal development.
Safety (metabolic tolerance) | At least daily during the first week of life, weekly up to 30 weeks postmenstrual age (when applicable), 30 weeks postmenstrual age (+-1d ), 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  Plasma and urinary urea (mg/dl), Plasma triglycerides (mg/dl), blood glucose (mg/dl)
Safety (haematology) | At least daily during the first week of life, weekly up to 30 weeks postmenstrual age (when applicable), 30 weeks postmenstrual age (+-1d ), 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  Complete blood count
Safety (gas-analysis) | At least daily during the first week of life, weekly up to 30 weeks postmenstrual age (when applicable), 30 weeks postmenstrual age (+-1d ), 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  Gas-analisys
Bone mineralisation | 6 weeks of age, 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  Plasma and urinary calcium and phosphorus, alkaline phosphatase, parathyroid hormone, osteocalcin measurements
Bone ultrasound (1) | 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  metacarpus speed of sound (m/s)
Bone ultrasound (2) | 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d )
  Metacarpus bone transmission time (ms)
Measurement of physical activity | 32 weeks postmenstrual age (+-1d ), 34 weeks postmenstrual age (+-1d ), 36 weeks postmenstrual age (+-1d ), 40 weeks postmenstrual age (+-1d) if still hospitalized
  Different levels of activity are assigned according to the Bruck's activity scale as described by Freymond et al. (24 hour continuous recording using a video camera). Levels of activity are defined as follows: 0, no body, arm, or leg movement, facial movement present or not with eyes closed or open; 1, arm or leg movement with eyes closed or open; 2, total body movement with eyes closed or open; 3, crying. Levels of activity in each group are expressed as percentage of time spent during the day in each level.
Morbidity | Hospital stay, on average 36 weeks postmenstrual age
  incidence of the main complication of prematurity
Mortality | hospital stay, on average 36 weeks postmenstrual age
  incidence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio P. Carnielli, MD, PhD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Ospedale G. Salesi, Ancona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Koletzko B, Goulet O, Hunt J, Krohn K, Shamir R; Parenteral Nutrition Guidelines Working Group; European Society for Clinical Nutrition and Metabolism; European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN); European Society of Paediatric Research (ESPR). 1. Guidelines on Paediatric Parenteral Nutrition of the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) and the European Society for Clinical Nutrition and Metabolism (ESPEN), Supported by the European Society of Paediatric Research (ESPR). J Pediatr Gastroenterol Nutr. 2005 Nov;41 Suppl 2:S1-87. doi: 10.1097/01.mpg.0000181841.07090.f4. No abstract available. PMID 16254497
- [Background] Embleton NE, Pang N, Cooke RJ. Postnatal malnutrition and growth retardation: an inevitable consequence of current recommendations in preterm infants? Pediatrics. 2001 Feb;107(2):270-3. doi: 10.1542/peds.107.2.270. PMID 11158457
- [Background] Burattini I, Bellagamba MP, Spagnoli C, D'Ascenzo R, Mazzoni N, Peretti A, Cogo PE, Carnielli VP; Marche Neonatal Network. Targeting 2.5 versus 4 g/kg/day of amino acids for extremely low birth weight infants: a randomized clinical trial. J Pediatr. 2013 Nov;163(5):1278-82.e1. doi: 10.1016/j.jpeds.2013.06.075. Epub 2013 Aug 12. PMID 23941670
- [Background] Bellagamba MP, Carmenati E, D'Ascenzo R, Malatesta M, Spagnoli C, Biagetti C, Burattini I, Carnielli VP. One Extra Gram of Protein to Preterm Infants From Birth to 1800 g: A Single-Blinded Randomized Clinical Trial. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):879-84. doi: 10.1097/MPG.0000000000000989. PMID 26418211
- [Background] Biolo G, Ciocchi B, Stulle M, Piccoli A, Lorenzon S, Dal Mas V, Barazzoni R, Zanetti M, Guarnieri G. Metabolic consequences of physical inactivity. J Ren Nutr. 2005 Jan;15(1):49-53. doi: 10.1053/j.jrn.2004.09.009. PMID 15648007
- [Background] Schulzke SM, Kaempfen S, Trachsel D, Patole SK. Physical activity programs for promoting bone mineralization and growth in preterm infants. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD005387. doi: 10.1002/14651858.CD005387.pub3. PMID 24752440
- [Result] Uthaya S, Thomas EL, Hamilton G, Dore CJ, Bell J, Modi N. Altered adiposity after extremely preterm birth. Pediatr Res. 2005 Feb;57(2):211-5. doi: 10.1203/01.PDR.0000148284.58934.1C. Epub 2004 Dec 20. PMID 15611357
- [Result] Prado CM, Heymsfield SB. Lean tissue imaging: a new era for nutritional assessment and intervention. JPEN J Parenter Enteral Nutr. 2014 Nov;38(8):940-53. doi: 10.1177/0148607114550189. Epub 2014 Sep 19. PMID 25239112
- [Result] Betto M, Gaio P, Ferrini I, De Terlizzi F, Zambolin M, Scattolin S, Pasinato A, Verlato G. Assessment of bone health in preterm infants through quantitative ultrasound and biochemical markers. J Matern Fetal Neonatal Med. 2014 Sep;27(13):1343-7. doi: 10.3109/14767058.2013.858317. Epub 2013 Nov 26. PMID 24215624